CLINICAL TRIAL: NCT02141113
Title: Double-Blind, Randomized, Placebo-Controlled, Single- Center, Dose Optimization Study Evaluating Efficacy and Safety of Guanfacine Hydrochloride in Combination With Psychostimulants in Adults Aged 18-65 Years With a Diagnosis of ADHD
Brief Title: Efficacy and Safety Eval of Guanfacine Hydrochloride in Combination With Psychostimulants in Adults (18-65).
Acronym: ADINT2012
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rochester Center for Behavioral Medicine (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1129704 ADINT
Record Dates: First submitted 2013-11-20; First posted 2014-05-19 (Estimated); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Adult Attention-Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guanfacine Hydrochloride (Active Comparator): 1. mg Guanfacine Hydrochloride (orally, QD)
  2. mg Guanfacine Hydrochloride (orally, QD)
  3. mg Guanfacine Hydrochloride (orally, QD)
  4. mg Guanfacine Hydrochloride (orally, QD)
  5. mg Guanfacine Hydrochloride (orally, QD)
  6. mg Guanfacine Hydrochloride (orally, QD)
  Interventions: Drug: Guanfacine Hydrochloride
- Sugar Pill (Placebo Comparator): 1. mg Placebo
  2. mg Placebo
  3. mg Placebo
  4. mg Placebo
  5. mg Placebo
  6. mg Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Guanfacine Hydrochloride — 1. mg Guanfacine Hydrochloride (orally)
  2. mg Guanfacine Hydrochloride (orally)
  3. mg Guanfacine Hydrochloride (orally)
  4. mg Guanfacine Hydrochloride (orally)
  5. mg Guanfacine Hydrochloride (orally)
  6. mg Guanfacine Hydrochloride (orally)
  Other Names: Intuniv
  Arms: Guanfacine Hydrochloride
Other: Placebo — Placebo of matching mg
  Arms: Sugar Pill

SUMMARY:
This is considered an investigator-initiated clinical research trial, which means that your study doctor is researching a particular medication (in this case a medication that is currently FDA- approved) for the treatment of AD/HD in individuals ages 6-17. The medication is guanfacine hydrochloride.

The hypothesis is that this medication could be used in adults with Attention Deficit/Hyperactivity Disorder who have not received satisfactory results with their current stimulant ADHD medication. The study drug is investigational for use in adults. Investigational means it has not been approved by the U.S. Food and Drug Administration (FDA) for use in adults.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether guanfacine hydrochloride used as an adjunct therapy (to subjects' current stimulant medication) would bring about a statistically significant improvement in AD/HD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male and females (non pregnant) ages 18-65
* Current diagnosis of ADHD and have met the DSM-IV-TR criteria for ADHD
* Currently taking an adequate dose stimulant to treat their ADHD (with a sub-optimal response). A suboptimal response is determined by a baseline score of 28 or greater on the ADHD-RS or a CGI score of 4 or greater.
* Subjects must be of normal intelligence
* English speaking
* Able to swallow pills.

Exclusion Criteria:

* Non pregnant or lactating females
* Severe Axis I and Axis II disorders
* Suicidal
* Tourette's
* Heart disease or any other serious chronic or acute unstable medical conditions/illnesses that would compromise participation or likely lead to hospitalization during the duration of the study.
* A known history or presence of cardiovascular, hepatic, renal, respiratory, or hematologic abnormalities, narrow angle glaucoma, or any other unstable medical or psychiatric conditions (as judged by the primary investigator)
* A current or recent history (within the past 6 months) of suspected substance abuse and/or drug dependence as defined by DSM-IV-TR criteria
* Healthy weight (not under or over as judged by investigator)
* No immediate family member of the investigator or research staff No involvement in a research study in the last 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-11; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel L Young, MD, Principal Investigator — Rochester Center for Behavioral Medicine
Locations (1):
- Rochester Center for Behavioral Medicine, Rochester Hills, Michigan, United States

REFERENCES:
- [Derived] Butterfield ME, Saal J, Young B, Young JL. Supplementary guanfacine hydrochloride as a treatment of attention deficit hyperactivity disorder in adults: A double blind, placebo-controlled study. Psychiatry Res. 2016 Feb 28;236:136-141. doi: 10.1016/j.psychres.2015.12.017. Epub 2015 Dec 17. PMID 26730446

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study site began recruiting for the trial in November 2012 and the last subject completed the final visit on 3/7/14. Recruitment was done from within the Rochester Center for Behavioral Medicine (a private mental health practice), as well as community outreach.
Pre-assignment Details: All participants were on a stable dose (as determined by the investigator) of a stimulant medication.
Groups:
- Guanfacine Hydrocholride; Sugar Pill Guanfacine Hydrocholride: 1. mg Guanfacine Hydrochloride (orally, QD)
  2. mg Guanfacine Hydrochloride (orally, QD)
  3. mg Guanfacine Hydrochloride (orally, QD)
  4. mg Guanfacine Hydrochloride (orally, QD)
  5. mg Guanfacine Hydrochloride (orally, QD)
  6. mg Guanfacine Hydrochloride (orally, QD)
  Guanfacine Hydrocholride: 1mg Guanfacine Hydrochloride (orally) 2mg Guanfacine Hydrochloride (orally) 3mg Guanfacine Hydrochloride (orally) 4mg Guanfacine Hydrochloride (orally) 5mg Guanfacine Hydrochloride (orally) 6mg Guanfacine Hydrochloride (orally)
Period: Overall Study
Arm/Group | Guanfacine Hydrocholride | Sugar Pill Guanfacine Hydrocholride
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guanfacine Hydrocholride | Sugar Pill Guanfacine Hydrocholride | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: ADHD-RS Change From Baseline to Endpoint
Description: The ADHD-RS is an 18-item scale based on DSM-IV criteria for ADHD. Each item is rated using a likert scale from 0 (none) to 3 (severe), with a total score range of 0-54, with higher scores indicating more symptoms/severity. In this study, we compared the mean change in ADHD-RS total score from baseline to endpoint of the study.
Time Frame: 0 weeks, 8 weeks
Population: All participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment: Guanfacine hydrochloride 1, 2, 3, 4, 5 or 6 mg
- Control Group: Matching placebo
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 13 | 13
units on a scale | 11.85 (7.63) | 10.92 (8.90)
Statistical Analysis 1: Comparison: Treatment vs Control Group; These scores were calculated by subtracting participants' endpoint scores from their initial baseline scores. These changed scores show the total change in ADHD symptoms over the course of the trial. Higher values indiicate improved functioning at the end of the trial compared to the beginning; Test type: Superiority or Other; p = .779, ANOVA

2. Secondary Outcome: The Clinical Global Impression (Severity)
Description: The Clinical Global Impression- Severity (CGI-S) is a clinician-assessed likert scale used to determine the severity of a patient's presenting symptoms. The scale evaluates a subject's illness from 1 (normal, not at all ill) to 7 (extremely ill). The results reported below indicate the magnitude of change in terms of mean points on a scale for each study condition (IMP or Placebo).
Time Frame: 0 weeks, 8 weeks
Population: Participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Placebo: Sugar pill guanfacine hydrochloride
Arm/Group | Guanfacine Hydrocholride | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale | .85 [.36 to 1.33] | 1.0 [.57 to 1.49]
Statistical Analysis 1: Comparison: Guanfacine Hydrocholride vs Placebo; Test type: Superiority; p = .834, ANOVA

3. Secondary Outcome: The Clinical Global Impression- Improvement (CGI-I)
Description: The Clinical Global Impression-Improvement (CGI-I) is a clinician-assessed likert scale measuring change in presenting symptoms from previous visit. The CGI-I is a 7-item scale with with 1 indicating that the subject has very much improved and 7 indicating that the subject has become very much worse.
Time Frame: 8 weeks
Population: Participants
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Guanfacine Hydrocholride: 1. mg Guanfacine Hydrochloride (orally, QD)
  2. mg Guanfacine Hydrochloride (orally, QD)
  3. mg Guanfacine Hydrochloride (orally, QD)
  4. mg Guanfacine Hydrochloride (orally, QD)
  5. mg Guanfacine Hydrochloride (orally, QD)
  6. mg Guanfacine Hydrochloride (orally, QD)
- Placebo: Sugar Pill Guanfacine Hydrocholride
Arm/Group | Guanfacine Hydrocholride | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale | 2.77 (1.01) | 2.92 (1.04)
Statistical Analysis 1: Comparison: Guanfacine Hydrocholride vs Placebo; Test type: Superiority or Other; p = .705, ANOVA

4. Other Pre Specified Outcome: Fatigue Symptoms Inventory (FSI) Change From Baseline to Endpoint
Description: The FSI is a 14-item self-report measure designed to assess the severity, frequency, and daily pattern of fatigue as well as its perceived interference with quality of life. Severity is measured on separate 11-point scales (0=not at all fatigued; 10=as fatigued as I could be) that assess most, least, and average fatigue since last visit, as well as current fatigue. The minimum score would be 0, maximum score would be 140. Scores below reflect mean improvement in FSI score from baseline (visit 0) to endpoint (visit 8). The FSI was used to measure safety and tolerability of study drug.
Time Frame: 0 weeks, 8 weeks
Population: Participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Guanfacine Hydrocholride | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale | 0.69 [-12.92 to 14.30] | 5.77 [-9.10 to 20.64]
Statistical Analysis 1: Comparison: Guanfacine Hydrocholride vs Placebo; Test type: Superiority or Other; p = .322, ANOVA

5. Other Pre Specified Outcome: Hamilton Anxiety Inventory Change From Baseline to Endpoint
Description: The Hamilton Anxiety Scale is a 14-items clinician-rated scale designed to measure anxiety severity. Each of the 14 items is scored from 0 (symptom not persent) to 4 (severe symptom). The total range is 0-56. A total score of less than 17 indicates mild severity, 18-24 indicates mild to moderate severity, and a score of 25-30 indicates moderate to severe symptoms. In this study, we compared the mean change in the Hamilton Anxiety scale from baseline to week 8 between guanfacine hyrdochloride and placebo-treated patients to assess safety and tolerability of study drug.
Time Frame: 0 weeks, 8 weeks
Population: Participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Guanfacine Hydrocholride | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale | 3.62 [.21 to 7.02] | 4.46 [1.49 to 7.44]
Statistical Analysis 1: Comparison: Guanfacine Hydrocholride vs Placebo; Test type: Superiority or Other; p = .043, ANOVA

6. Other Pre Specified Outcome: Arizona Sexual Experiences Scale (ASEX) Change From Baseline to Endpoint
Description: The Arizona Sexual Experiences Scale (ASEX) is both a self-administered or clinician-administered questionnaire. It is a user-friendly 5-item rating scale. The ASEX utilizes short, easy to understand, and less intrusive questions that explores the follwoing aspects of sexuality:
  1. sex drive
  2. arousal 3a. penile erection 3b. vaginal lubrication
  4. ability to reach orgasm 5. satisfaction from orgasm Scores can range from a minimum of 6 (indicating minimal problems with sexual functioning) to 36 (indicating maximum problems with sexual functioning).
  Mean change from baseline (visit 0) to endpoint (visit 8) are presented below. The ASEX was used to assess safety and tolerability of drug from baseline to endpoint
Time Frame: 0 weeks, 8 weeks
Population: All participants were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Treatment Group: Guanfacine Hydrochloride 1, 2, 3, 4, 5, or 6 mg
- Placebo: guanfacine hydrochloride sugar pill
Arm/Group | Treatment Group | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale | -.77 [-2.21 to 0.67] | 1.31 [-1.91 to 4.53]
Statistical Analysis 1: Comparison: Treatment Group vs Placebo; Test type: Superiority or Other; p = .212, ANOVA

7. Other Pre Specified Outcome: Hamilton Depression Rating Scale (HAM-D) Change From Baseline to Endpoint
Description: The HAM-D is a clinician administered multiple item scale used to provide an indication of depression symptom severity. It is designed for adults. Each item on the questionnaire is scored on a 3 or 5 point scale. The HAM-D is comprised of 21 items, however, the total score is based on the sum of the scores from the first 17 items. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. Thus the possible total score range is 0 (minimum) to 40 (maximum) with a higher score indicating greater severity of depression. Accordingly, a low HAM-D score would indicate a better outcome. Mean change scores from baseline (visit 0) to endpoint (visit 8) are presented below.
Time Frame: 0 weeks, 8 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Guanfacine Hydrocholride | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale | 3.31 [.14 to 6.48] | 4.23 [1.93 to 6.53]

8. Other Pre Specified Outcome: The Pittsburgh Sleep Quality Index (PSQI) Change From Baseline to Endpoint
Description: The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep by measuring seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. The individual self rates each of these seven areas of sleep. Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale. Total score range is from 0 to 21. The mean improvement from baseline (visit 0) to endpoint (visit 8) are presented below. PSQI was used to assess safety and tolerability of study drug.
Time Frame: 0 weeks, 8 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Guanfacine Hydrocholride | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale | 2.69 [-1.24 to 6.63] | 2.08 [-0.01 to 4.16]

ADVERSE EVENTS:
Groups:
- Control Group: Placebo 1, 2, 3, 4, 5, or 6 mg
Arm/Group | Treatment Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
Relatively small sample size and herterogenous sample (male paticipants = 14 and female participants = 12).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No